CLINICAL TRIAL: NCT02338128
Title: The Cardiovascular Protective Effects of Febuxostat in Peritoneal Dialysis Patients: a Prospective Cohort Study
Brief Title: The Cardiovascular Protective Effects of Febuxostat in Peritoneal Dialysis Patients
Status: Completed | Type: Observational
Sponsor: Shanghai 10th People's Hospital (Other)
Responsible Party: Principal Investigator, Ai Peng, Chief of department of Nephrology & Rheumatology, Shanghai 10th People's Hospital
Other Study IDs: FPD2015
Record Dates: First submitted 2015-01-09; First posted 2015-01-14 (Estimated); Last update posted 2019-07-24 (Actual); Status verified 2019-07

CONDITIONS: Disorders Associated With Peritoneal Dialysis; Hyperuricemia
Keywords: peritoneal dialysis; hyperuricemia; cardiovascular; Febuxostat
MeSH Terms: conditions — Hyperuricemia

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: Yes

SUMMARY:
The purpose of this study is to determine whether Febuxostat could protect cardiovascular function of peritoneal dialysis patients by lowering serum uric acid.

DETAILED DESCRIPTION:
Patients with more than 3-month-history of peritoneal dialysis and hyperuricemia. Use Febuxostat to control their serum uric acid for 1 year. To observe the cardiovascular events of patients, and compare and evaluate the changes of heart function, heart construction, serum cardiac markers and brain natriuretic peptide (BNP) levels before and after Febuxostat treatment.

ELIGIBILITY:
Inclusion Criteria:

- Peritoneal dialysis for more than 3 months with hyperuricemia.

Exclusion Criteria:

1. Acute hepatopathy or liver dysfunction (Aspartate transaminase and/or alanine aminotransferase exceed 2 times of normal range)
2. Heart failure (stage IV, NYHA), unstable angina, acute stroke
3. Severe lung disease or cancer
4. unable to sign the informed consent form or disagree following-up.

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Peritoneal dialysis patients with hyperuricemia
Sampling Method: Non-Probability Sample
Enrollment: 50 (Actual)
Dates: Start 2015-01; Primary Completion 2018-01 (Actual); Study Completion 2018-01 (Actual)

PRIMARY OUTCOMES:
cardiovascular events (heart failure, myocardial infarction, unstable angina which need hospitalization，heart surgery, or death caused by cardiovascular disease.) | 1 year
  heart failure, myocardial infarction, unstable angina which need hospitalization，heart surgery, or death caused by cardiovascular disease.

SECONDARY OUTCOMES:
Serum uric acid | 1st month, 2nd month, 3rd month, 6th month, 9th month, 12th month
  blood test for serum uric acid
cardiovascular function (Heart construction and cardiac ejection fraction determined by echocardiography; blood test: cardiac markers including troponin,myoglobin and creatinine kinase, MB isoenzyme (CK-MB), brain natriuretic peptide) | 6 months
  Heart construction and cardiac ejection fraction determined by echocardiography; blood test: cardiac markers including troponin,myoglobin and creatinine kinase, MB isoenzyme (CK-MB), brain natriuretic peptide.

CONTACTS AND LOCATIONS:
Overall Officials: Ling Wang, MD, PhD, Study Chair — Department of Nephrology & Rheumatology, Shanghai Tenth People's Hospital
Locations (1):
- Department of Nephrology & Rheumatology, Shanghai Tenth People's Hospital, Shanghai, Shanghai Municipality, China